CLINICAL TRIAL: NCT03149835
Title: Acute Non-invasive Ventilation Reduces Cerebral Blood Flow in COPD Patients and Healthy Controls Without Effects on Cognitive Function
Brief Title: NIV Reduces CBF in COPD Patients Without Cognitive Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Ceara (Other)
Responsible Party: Principal Investigator, Marcelo Alcantara Holanda, MD, PhD, Universidade Federal do Ceara
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 021.04.07
Record Dates: First submitted 2017-05-02; First posted 2017-05-11 (Actual); Last update posted 2017-05-11 (Actual); Status verified 2007-04

CONDITIONS: COPD; Non-invasive Ventilation; Cognitive Impairment; Cerebral Blood Flow
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Cognitive Dysfunction | interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COPD (Experimental): After study enrollment, 15 days before the performance of the experimental protocol, patients performed neurocognitive tests (Digit Span Test, Digit Symbol-Coding, Corsi Block-tapping, Trail Making Test A and B and Stroop Test) and NIV adaptation. Pulmonary function (spirometry) was measured in all subjects after a thorough medical history and physical examination. Before initiating the protocol, patients were asked about discomfort related to NIV or any aspect of the experiment.
  CBF was measured by transcranial Doppler by mean of LMCAFV immediately before NIV, during NIV at 5, 30 and 60 minutes and after NIV removal at 5 and 30 minutes. ABG were collected immediately before the experiment, after one hour of NIV breathing and 30 minutes after NIV discontinuation.
  Interventions: Other: Non-invasive ventilation
- Healthy Control (Experimental): After study enrollment, 15 days before the performance of the experimental protocol, patients performed neurocognitive tests (Digit Span Test, Digit Symbol-Coding, Corsi Block-tapping, Trail Making Test A and B and Stroop Test) and NIV adaptation. Pulmonary function (spirometry) was measured in all subjects after a thorough medical history and physical examination.
  CBF was measured by transcranial Doppler by mean of LMCAFV immediately before NIV, during NIV at 5, 30 and 60 minutes and after NIV removal at 5 and 30 minutes. ABG were collected immediately before the experiment, after one hour of NIV breathing and 30 minutes after NIV discontinuation.
  Interventions: Other: Non-invasive ventilation

INTERVENTIONS:
Other: Non-invasive ventilation — NIV was provided by BiPAP-Vision™ ventilator (Philips Respironics Inc, Murrysville, PA, USA) set at the BIPAP mode and applied by a nasal mask, with room air, for 60 minutes. Volunteers were studied during the application of NIV (inspiratory pressure of 14cmH2O and expiratory pressure of 4cmH2O), with a pressure support of 10cmH2O and without oxygen support (FIO2 0.21). These pressure levels were chosen based on the current practice of NIV in the intensive care setting.

SUMMARY:
Objectives: Investigate the acute NIV effects on CBF and cognitive functions in COPD patients. Methods: Nine non-hypercapnic stable COPD subjects (FEV1/FVC < lower limit of normal) and twelve healthy controls were enrolled. CBF (transcranial Doppler), cognitive functions, respiratory and cardiovascular response were tested at baseline, during and after non-invasive ventilation.

DETAILED DESCRIPTION:
Nine COPD patients were screened from the Respiration Laboratory (RespLab) of Federal University of Ceará, and twelve sedentary controls from the general population were also assessed. All patients were under stable medical treatment at least two months, and COPD diagnosis was made according to GOLD guidelines. Patients were excluded if they had heart disease, arterial hypertension, other debilitating pulmonary or non-pulmonary diseases, depression, preexisting psychiatric or neurologic disorders, stroke, motor impairment, visual or hearing disabilities, mini-mental scale examination score below 20 points, and any disease that could influence the effectiveness of NIV application or the performance of cognitive tests. The control group consisted of healthy and nonsmoking volunteers.

After study enrollment, 15 days before the performance of the experimental protocol, patients performed neurocognitive tests (Digit Span Test, Digit Symbol-Coding, Corsi Block-tapping, Trail Making Test A and B and Stroop Test) and NIV adaptation. Pulmonary function (spirometry) was measured in all subjects after a thorough medical history and physical examination. Before initiating the protocol, patients were asked about discomfort related to NIV or any aspect of the experiment. CBF, capnometry, arterial blood gases (ABG) and neurocognitive tests were performed before, during and after NIV.

CBF was measured by transcranial Doppler by mean of LMCAFV immediately before NIV, during NIV at 5, 30 and 60 minutes and after NIV removal at 5 and 30 minutes. ABG were collected immediately before the experiment, after one hour of NIV breathing and 30 minutes after NIV discontinuation. Respiratory rate (RR), tidal volume (VT), oxygen saturation by pulse oximetry (SpO2), heart rate (HR), minute ventilation (VE) and mean systemic arterial blood pressure (MAP) were continuously measured by a multiparameter monitor (Dixtal DX-2010™, Dixtal, Manaus, Brazil) both on spontaneous respiration and NIV.

Subjects were tested in the morning and investigated while awake and at the supine position, throughout the experiment.

ELIGIBILITY:
Inclusion Criteria:

* All patients were under stable medical treatment at least two months
* COPD diagnosis was made according to GOLD guidelines

Exclusion Criteria:

* heart disease, arterial hypertension, other debilitating pulmonary or non-pulmonary diseases, depression, preexisting psychiatric or neurologic disorders, stroke, motor impairment, visual or hearing disabilities, mini-mental scale examination score bellow 20 points, and any disease that could influence the effectiveness of NIV application or the performance of cognitive tests

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-05-01 (Actual); Primary Completion 2011-05-01 (Actual); Study Completion 2011-05-31 (Actual)

PRIMARY OUTCOMES:
Cognitive Function | Neurocognitive tests were applied after 60 min of NIV
  Change from baseline in a neuropsychological test was performed after 60 min of NIV to evaluate cognitive dysfunction.

SECONDARY OUTCOMES:
Cerebral blood flow | Cerebral blood flow were tested after 60 min of NIV
  A 2 MHz pulsed Transcranial Doppler (TCD) ultrasound Doppler-boxTM DLWTM Doppler system device (Compumedics DLWTM Doppler Company, Germany) was used to measure the change from baseline on left MCAFV (LMCAFV).
  The ultrasound probe was placed over the left temporal bone, just above the zygomatic arch (temporal window) to obtain LMCAF.

IPD SHARING:
Plan to Share IPD: No